CLINICAL TRIAL: NCT05866900
Title: The Impact of Daily CarboHydrate Intake on Glycemic Control in Children and Adolescents With Type 1 Diabetes Using an Advanced Hybrid Closed-loop System (Medtronic MiniMed 780G): a Multi-center Real-world Observational Study
Brief Title: The Impact of Daily Carbohydrate Intake on Glycemic Control in Children and Adolescents With Type 1 Diabetes Using an Advanced Hybrid Closed-loop System
Acronym: CHOco-AID
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Ljubljana, Faculty of Medicine (Other)
Collaborators: University of Messina (Other)
Responsible Party: Sponsor
Other Study IDs: CHOco-AID
Record Dates: First submitted 2023-05-10; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: MiniMed 780G; automated insulin delivery; nutrition; diet; time in range; insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: MiniMed 780G with SmartGuard activated — The MiniMed 780G system consists of a MiniMed 780G Insulin Pump connected to Guardian 4 Sensor or Guardian 3 Sensor, using an automated insulin delivery algorithm called SmartGuard.

SUMMARY:
Lifestyle factors, including diet, play an important role in the achievement of glycemic targets in patients with diabetes, even with the use of automated insulin delivery (AID) systems. Advanced hybrid closed-loop systems (AHCL), by implementing innovative and powerful control algorithms, have been shown to improve the post-meal glycemic control in their users through the delivery of automatic correction boluses. However, data about the influence of the daily amount of carbohydrate intake on glycemic outcomes in youth with type 1 diabetes using AHCL are missing. Therefore, this study will evaluate the association between daily carbohydrate intakes and meal patterns on glycemic control of young people living with type 1 diabetes using an AHCL system (Medtronic MiniMed 780G; Medtronic, Northridge, California) under real-life conditions.

ELIGIBILITY:
Inclusion Criteria:

* Patients with type 1 diabetes
* Patients aged 7-18 years
* Patients using Medtronic MiniMed 780G with SmartGuard activated
* Patients whose informed consent has been obtained
* >70% CGM data during observational period

Exclusion Criteria:

* Patients with partial clinical remission according to the Hvidovre Study Group definition
* Concomitant treatment with steroids or other drugs known to interfere with blood glucose levels
* Previous diagnosis of psychological or eating disorders

Ages: 7 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: Participants will be recruited from electronical records of two Pediatric Diabetes departments located in Slovenia and Italy
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2023-05-15 (Estimated); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Time in range (%) | 6 months
  Time spent with sensor glucose between 70 and 180 mg/dl (3.9 and 10 mmol/L)
Time above range level 1 (%) | 6 months
  Time spent with sensor glucose between 180 and 250 mg/dl (10.1 and 13.9 mmol/L)
Time above range level 2 (%) | 6 months
  Time spent with sensor glucose > 250 mg/dl (13.9 mmol/L)
Time below range level 1 (%) | 6 months
  Time spent with sensor glucose between 54 and 70 mg/dl (3.0 and 3.8 mmol/L)
Time below range level 2 (%) | 6 months
  Time spent with sensor glucose < 54 mg/dl (3.0 mmol/L)
Mean sensor glucose (mg/dl or mmol/L) | 6 months
Coefficient of variation (%) | 6 months

SECONDARY OUTCOMES:
BMI Z-score | Baseline, 3 months, 6 months
Weight Z-score | Baseline, 3 months, 6 months
Height Z-score | Baseline, 3 months, 6 months

IPD SHARING:
Plan to Share IPD: Undecided